CLINICAL TRIAL: NCT07299110
Title: Effect of Whey Protein Versus Egg Albumen Protein Challenge on Blood Ammonia Level in Patients of Decompensated Ethanol Related Cirrhosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-74
Record Dates: First submitted 2025-07-31; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Decompensated Cirrhosis Ethanol Related
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- whey protein and egg albumen (Experimental): Each participant will receive two oral protein challenges in a crossover design:
  1. Whey Protein Challenge: 30g of whey protein in 200-250 mL water on Day 1
  2. Egg Albumen Challenge: 30g of egg albumen protein in 200-250 mL water on Day 2
  Interventions: Dietary Supplement: Whey Protein; Dietary Supplement: Egg Albumen

INTERVENTIONS:
Dietary Supplement: Whey Protein — Whey Protein Challenge: 30g of whey protein in 200-250 mL water on Day 1.
Dietary Supplement: Egg Albumen — Egg Albumen Challenge: 30g of egg albumen protein in 200-250 mL water on Day 2.

SUMMARY:
In cirrhosis, altered nitrogen metabolism and reduced hepatic clearance of ammonia contribute to the development of Minimal Hepatic Encephalopathy (MHE)-a subclinical but functionally debilitating condition. While adequate protein intake is essential to prevent sarcopenia in cirrhotic patients, the type of protein consumed can significantly influence postprandial ammonia generation, thereby affecting neurocognitive status.

This study investigates the differential ammoniagenic potential of two commonly used high-protein nutritional supplements-Whey protein, which is rich in branched-chain amino acids (BCAAs) and rapidly absorbed, and egg albumen protein, which is slower digesting and higher in aromatic amino acids (AAAs), potentially more ammoniagenic.

In a crossover pilot design, 50 patients with decompensated ethanol-related cirrhosis will undergo two separate standardized protein challenges with 30g of each protein, spaced 24 hours apart. Venous ammonia levels and MHE parameters (via PHES/Stroop test) will be recorded pre- and 3 hours post-challenge.

The primary objective is to compare the change in blood ammonia between the two protein types. Secondary objectives include assessing MHE induction or worsening, and analysing the correlation between ammonia changes and cognitive decline.

By directly comparing the metabolic and neurocognitive response to distinct protein sources, this study will help inform safer dietary practices and refine nutritional supplementation in cirrhosis, especially for those at risk of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Known or newly diagnosed (clinical, imaging) case of decompensated ethanol related cirrhosis patients.
2. Age (18-70 years).
3. Informed consent to participate in the study.

Exclusion Criteria:

1. History of overt HE (West Haven grade II or more).
2. Last Intake <1.5 months.
3. CKD (creatinine >1.5 mg/dL), active infection, GI bleeding in past 2 weeks.
4. Severe anaemia (Hb <7 g/dL) or hypoalbuminemia (<2.0 g/dL).
5. Known egg or dairy allergy.
6. Those on sedatives, antidepressant or anti-psychiatric medication.
7. Unable to understand the language or instructions.
8. Hepatocellular Carcinoma.
9. TIPS.
10. Receiving rifaximin or lactulose.
11. Diarrhea, SIBO or malabsorptive syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the effects of whey protein versus egg albumen protein oral challenge in blood ammonia level after 3 hours in decompensated ethanol related cirrhosis. | 24 hours

SECONDARY OUTCOMES:
To determine the prevalence of minimal hepatic encephalopathy (MHE). | 24 hours
To compare the prevalence of MHE in 24 hours following whey protein versus egg albumen protein challenge. | 24 hours
Initial lab parameters that predict protein challenge induced MHE. | 24 hours
Number of participants with treatment related adverse effects accessed by CTCAE v4.0 | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institiute of liver and biliary sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided